CLINICAL TRIAL: NCT04913363
Title: The Emotional, Physical and Cognitive Benefits of Purposeful Green Space Activities on Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Jennifer Roe, Professor, University of Virginia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSR210100; UL1TR003015 (NIH)
Record Dates: First submitted 2021-05-10; First posted 2021-06-04 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Loneliness; Social Isolation; Mood; Well Aging; Physical Activity; Mobility Limitation
MeSH Terms: conditions — Social Isolation; Motor Activity; Mobility Limitation | interventions — Parks, Recreational

STUDY DESIGN:
Intervention Model Description: The study was designed in a single group, where participants will be complete the interventions (green space activities) in this order: Citizen Science, Walking, Planting. However, participants may or may not show up on the day of an activity. i.e. participants may skip one or more interventions, even though that was not the intent of the study design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Walking (Experimental): This contemplative activity will see users taken to a local green space area near their center and encouraged to walk around the space. It is anticipated walks will last around 15-20 minutes.
  Interventions: Other: Green space
- Citizen Science (Experimental): This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Interventions: Other: Green space
- Planting (Experimental): This physical activity will see users, lead by a local Master Gardener, engage with planting vegetables/fruit in raised beds. Not only will this allow users a chance to engage physically with nature, but it is anticipated that the grown produce will be used for center users.
  Interventions: Other: Green space

INTERVENTIONS:
Other: Green space — Green space in which activities take place

SUMMARY:
This project explores if various nature based activities can lead to acute improvements in emotional, physical and cognitive health outcomes and encouraging senior center (JABA) service users to return to a safe environment. The activities the investigators will use include walking in nature, engaging in physical planting and cerebral, citizen science based activities.

DETAILED DESCRIPTION:
This study builds on the previous experimental work and expands it to focus on older adults in the Charlottesville area. The study objective is to understand the impact of different types of activities in green settings on physical and mental health outcomes in older adults at JABA centers using a repeated measures, crossover design in 20 participants.

There are three activity sessions in this project; walking (contemplative), planting (physical) and citizen science (cerebral). The walking condition will be a short green walk (10-15 minutes). The planting session will be run by JABA staff and a Master Gardener and will allow participants an opportunity to be outdoors and plant and tend to plants. The citizen science session will be run by JABA staff and a consultant and will rely less on physical exertion but rather focus on understanding green space at a more academic level. All sessions will be outdoors and will follow COVID-19 guidelines in place at the time of testing.

Outcome Measures The investigators will use various measures to assess the impact of green activity on emotional, physical and cognitive health outcomes, including;

* Loneliness; measured by the UCLA Loneliness Scale, a 3-item scale that captures feelings of loneliness.
* Belonging; measured by the General Belonging Scale (GBS), a 12-item scale capturing social acceptance/inclusion and social rejection/exclusion.
* Acute Mood; pre and post measures of mood will be taken using the UWIST Mood Adjective Checklist (MACL), an acute measure of hedonic tone, stress and arousal.
* Restoration; Psychological restorative qualities of the setting measured by the Perceived Restorativeness Scale, a three point scale determining the restorative quality of activity spaces.
* Physical Activity_OMNIT; In addition to the arousal measure of the MACL, the investigators used the 11 point scale (from 0 to 10) of the OMNIT Perceived Exertion scale (tiredness), to understand how physically tired the activities made them.
* Physical Activity_OMNIH; In addition to the arousal measure of the MACL, the investigators used the 11 point scale (from 0 to 10) of the OMNIH Perceived Exertion scale (exertion), to understand how much perceived physical effort participants put in.
* Accelerometer; the investigators will use accelerometers to measure participant movement throughout the activities to correlate with physical activity measures.

All outcome measures will be scored and subsequently analysed using a one-way ANOVA to determine if experimental condition leads to any statistically significant difference between outcome scores. The investigators will look for correlations between outcome measures in order to establish relationships between variables.

The investigators will also send a short survey to a number of JABA service users (n=30) to understand mood, wellbeing and current barriers to returning to their local JABA center. This survey will include the UCLA Loneliness Scale, the GBS, mood and physical activity measures included above, as well as broader questions assessing their experience of the lockdown and their needs for safe return to the center.

Participants will be sent consent information in advance and have an opportunity to talk to the research time prior to attending their first session. For all conditions, participants would meet at a pre-determined location near their local JABA center and taken to the activity site directly. Participants will complete the short surveys, listed above, both pre and post their activity. All activities will last around 20 minutes. Participants will return for two consecutive weeks to undertake the alternative activities to which they originally completed.

Activities Participants will undertake three activities, on separate days, throughout this project.

1. Walking; this contemplative activity will see users taken to a local green space area near their center and encouraged to walk around the space. It is anticipated that walks will last around 15-20 minutes.
2. Planting; this physical activity will see users, lead by a local Master Gardener, engage with planting vegetables/fruit in raised beds. Not only will this allow users a chance to engage physically with nature, but it is anticipated that the grown produce will be used for center users.
3. Citizen Science; this cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years
* A JABA center user
* Can walk unassisted for 20 minutes
* Willing to comply with COVID-19 regulations

Exclusion Criteria:

* Under 65 years
* Never used a JABA center
* unable to walk unassisted for 20 minutes.
* Unwilling to comply with COVID-19 regulations

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2022-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Roe, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Citizen Science + Walking + Planting: Participants who completed all three interventions, in this order.
  Citizen Science: This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Walking: This contemplative activity will see users taken to a local green space area near their center and encouraged to walk around the space. It is anticipated walks will last around 15-20 minutes.
  Planting: This physical activity will see users, lead by a local Master Gardener, engage with planting vegetables/fruit in raised beds. Not only will this allow users a chance to engage physically with nature, but it is anticipated that the grown produce will be used for center users.
  Green space: Green space in which activities take place
- Citizen Science + Walking: Participants who completed Citizen Science + Walking, in this order.
  Citizen Science: This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Walking: This contemplative activity will see users taken to a local green space area near their center and encouraged to walk around the space. It is anticipated walks will last around 15-20 minutes.
  Green space: Green space in which activities take place
- Citizen Science + Planting: Participants who completed Citizen Science and Planting, in this order.
  Citizen Science: This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Planting: This physical activity will see users, lead by a local Master Gardener, engage with planting vegetables/fruit in raised beds. Not only will this allow users a chance to engage physically with nature, but it is anticipated that the grown produce will be used for center users.
  Green space: Green space in which activities take place
- Citizen Science: Participants completed Citizen Science only.
  Citizen Science: This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Green space: Green space in which activities take place.
- Walking: Participants Complete Walking Only
  Walking: This contemplative activity will see users taken to a local green space area near their center and encouraged to walk around the space. It is anticipated walks will last around 15-20 minutes.
  Green space: Green space in which activities take place
- Planting: Participants completed Planting only.
  Planting: This physical activity will see users, lead by a local Master Gardener, engage with planting vegetables/fruit in raised beds. Not only will this allow users a chance to engage physically with nature, but it is anticipated that the grown produce will be used for center users.
  Green space: Green space in which activities take place
Period: Overall Study
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Started | 12 | 1 | 1 | 3 | 5 | 2
Completed | 12 | 1 | 1 | 3 | 5 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Citizen Science + Walking + Planting: Participants who completed all three interventions.
  Citizen Science: This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Walking: This contemplative activity will see users taken to a local green space area near their center and encouraged to walk around the space. It is anticipated walks will last around 15-20 minutes.
  Planting: This physical activity will see users, lead by a local Master Gardener, engage with planting vegetables/fruit in raised beds. Not only will this allow users a chance to engage physically with nature, but it is anticipated that the grown produce will be used for center users.
  Green space: Green space in which activities take place
- Citizen Science + Walking: Participants who completed Citizen Science + Walking
  Citizen Science: This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Walking: This contemplative activity will see users taken to a local green space area near their center and encouraged to walk around the space. It is anticipated walks will last around 15-20 minutes.
  Green space: Green space in which activities take place
- Citizen Science + Planting: Participants who completed Citizen Science and Planting.
  Citizen Science: This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Planting: This physical activity will see users, lead by a local Master Gardener, engage with planting vegetables/fruit in raised beds. Not only will this allow users a chance to engage physically with nature, but it is anticipated that the grown produce will be used for center users.
  Green space: Green space in which activities take place
- Total: Total of all reporting groups
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting | Total
Number analyzed (Participants) | 12 | 1 | 1 | 3 | 5 | 2 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 12 | 1 | 1 | 3 | 5 | 2 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.16 (2.85) | 74.0 (0) | 72 (0) | 78.3 (3.29) | 74 (.63) | 75 (9) | 72.62 (4.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 1 | 3 | 2 | 1 | 16
  Male | 4 | 0 | 0 | 0 | 3 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 1 | 1 | 2 | 4 | 1 | 19
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 1 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 0 | 1 | 3
  White | 12 | 1 | 1 | 1 | 5 | 1 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 1 | 1 | 3 | 5 | 2 | 24

OUTCOME MEASURES:

1. Primary Outcome: Loneliness (Time 1)
Description: Loneliness was measured by the University of California, Los Angeles (UCLA) Loneliness Scale, a 3-item scale that captures feelings of loneliness. Scores range from 3 to 9 with higher scores indicating higher levels of perceived loneliness
Time Frame: Pre activity
Population: Only 2 (of 3) participants from the Citizen Science group completed the UCLA scale.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Citizen Science + Walking + Planting: Participants who completed all three interventions.
  Citizen Science: This cerebral activity sees users engage with local green spaces, under the instruction of a citizen scientist, to learn about the intricacies of the space. This may include lichen counts (or similar) where the main outcome is learning based.
  Walking: This contemplative activity will see users taken to a local green space area near their center and encouraged to walk around the space. It is anticipated walks will last around 15-20 minutes.
  Planting: This physical activity will see users, lead by a local Master Gardener, engage with planting vegetables/fruit in raised beds. Not only will this allow users a chance to engage physically with nature, but it is anticipated that the grown produce will be used for center users.
  Green space: Green space in which activities take placece in which activities take place
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 12 | 1 | 1 | 2 | 5 | 2
units on a scale | 4.08 (1.084) | 5 (0) | 3 (0) | 3 (0) | 3.6 (0.894) | 3 (0)

2. Primary Outcome: Loneliness (Time 2)
Description: as for outcome 1
Time Frame: Post activity (20 minutes after pre-activity measure)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 12 | 1 | 1 | 3 | 5 | 2
units on a scale | 4.25 (1.357) | 5 (0) | 3 (0) | 4.33 (2.309) | 3.4 (0.894) | 3 (0)

3. Primary Outcome: Social Isolation (Time 1)
Description: Social Isolation was measured by the General Belonging Scale (GBS), a 12-item scale capturing social acceptance/inclusion and social rejection/exclusion. Scores will range from 12 to 84, with higher scores indicating higher levels of perceived belonging.
Time Frame: Pre activity
Population: Only 2 (of 3) participants from the Citizen Science group completed the GBS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 12 | 1 | 1 | 2 | 5 | 2
units on a scale | 71.42 (12.894) | 56 (0) | 83 (0) | 74 (2.828) | 70.4 (13.24) | 79 (7.071)

4. Primary Outcome: Social Isolation (Time 2)
Description: as for outcome 3
Time Frame: Post activity (20 minutes after pre-activity measure)
Population: Only 4 (of 5) participants from the Walking group completed the GBS measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 12 | 1 | 1 | 3 | 4 | 2
units on a scale | 72.18 (13.121) | 51 (0) | 84 (0) | 65 (4.583) | 67.75 (17.481) | 79.5 (6.364)

5. Primary Outcome: Mood_hedonic Tone (Time 1)
Description: Pre measures of mood (hedonic tone) was taken using the University of Wales Institute of Science and Technology (UWIST) Mood Adjective Checklist (MACL), an average measure of hedonic tone. The subscale will range from 4 to 16, with higher scores indicating higher valence.
Time Frame: Pre activity
Population: For the Citizen Science group, only 2 (of 3) participants completed the measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 12 | 1 | 1 | 2 | 5 | 2
units on a scale | 14.92 (1.975) | 14 (0) | 16 (0) | 12.5 (0.707) | 13.6 (2.191) | 14 (2.828)

6. Primary Outcome: Mood_hedonic Tone (Time 2)
Description: Post measures of (hedonic tone) was taken using the University of Wales Institute of Science and Technology (UWIST) Mood Adjective Checklist (MACL), an average measure of hedonic tone. The subscale will range from 4 to 16, with higher scores indicating higher valence.
Time Frame: Post activity (20 minutes after pre-activity measure)
Population: For the CS+Walking+Planting group, only 11 (of 12) participants completed the measure. For the Citizen Science group, only 2 (of 3) participants completed the measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 11 | 1 | 1 | 2 | 5 | 2
units on a scale | 15.27 (1.489) | 16 (0) | 16 (0) | 14.5 (2.121) | 15.2 (1.304) | 14.5 (2.121)

7. Primary Outcome: Well Aging_ Using Perceived Restorativeness Scale
Description: Psychological restorative qualities of the setting was measured by the Perceived Restorativeness Scale, a three point scale determining the restorative quality of activity spaces. Scores range from 4 to 28, with higher scores indicating higher levels of perceived restoration.
Time Frame: Post activity (20 minutes after pre-activity measure). This measure is a post-condition measure only that measures restoration as a result of the condition. This cannot be done before exposure to the condition.
Population: For the CS+Walking+Planting group, only 11 (of 12) participants completed the measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 11 | 1 | 1 | 3 | 5 | 2
units on a scale | 26.55 (2.207) | 24 (0) | 28 (0) | 24.67 (3.512) | 25.4 (2.881) | 27 (0)

8. Primary Outcome: Physical Activity_OMNIT
Description: In addition to the arousal measure of the MACL, the investigators used the 11 point scale (from 0 to 10) of the OMNIT Perceived Exertion scale (tiredness), to understand how physically tired the activities made them. Lower scores indicate the tasks are easy; higher scores indicate the tasks are hard.
Time Frame: Post activity (20 minutes after pre-activity measure). OMNIT is administered post-activity ONLY.
Population: For the CS+Walking+Planting group, only 11 (of 12) participants completed the measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 11 | 1 | 1 | 3 | 5 | 2
units on a scale | 0.73 (0.786) | 5 (0) | 0 (0) | 0.67 (0.577) | 1.2 (1.095) | 0.5 (0.707)

9. Primary Outcome: Physical Activity_OMNIH
Description: In addition to the arousal measure of the MACL, the investigators used the 11 point scale (from 0 to 10) of the OMNIH Perceived Exertion scale (exertion), to understand how much perceived physical effort participants put in. Lower scores indicate the tasks are easy; higher scores indicate the tasks are hard.
Time Frame: Post activity (20 minutes after pre-activity measure). OMNIH is administered post-activity ONLY.
Population: For the CS+Walking+Planting group, only 11 (of 12) participants completed the measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 11 | 1 | 1 | 3 | 5 | 2
units on a scale | 0.91 (0.944) | 6 (0) | 2 (0) | 1 (0) | 1.6 (1.14) | 1.5 (0.707)

10. Primary Outcome: Mood_Stress (Time 1)
Description: Pre measures of mood (stress) was taken using the University of Wales Institute of Science and Technology (UWIST) Mood Adjective Checklist (MACL), an average measure of stress. The subscale will range from 4 to 16, with higher scores indicating higher stress.
Time Frame: Pre activity
Population: For the Citizen Science group,, only 2 (of 3) participants completed the measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 12 | 1 | 1 | 2 | 5 | 2
units on a scale | 5.42 (2.065) | 11 (0) | 4 (0) | 4 (0) | 7.6 (4.099) | 7 (4.243)

11. Primary Outcome: Mood_Stress (Time 2)
Description: Post measures of mood (stress) was taken using the University of Wales Institute of Science and Technology (UWIST) Mood Adjective Checklist (MACL), an average measure of stress. The subscale will range from 4 to 16, with higher scores indicating higher stress.
Time Frame: Post activity (20 minutes after pre-activity measure)
Population: For the CS+Walking+Planting group, only 11 (of 12) participants completed the measure. For the CS group, only 2 (of 3) participants completed the measure..
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 11 | 1 | 1 | 2 | 5 | 2
units on a scale | 4.55 (1.036) | 4 (0) | 4 (0) | 4 (0) | 5.2 (1.789) | 5.5 (2.121)

12. Primary Outcome: Mood_arousal (Time 1)
Description: Pre measures of mood (arousal) was taken using the University of Wales Institute of Science and Technology (UWIST) Mood Adjective Checklist (MACL), an average measure of arousal. The subscale will range from 4 to 16, with higher scores indicating higher arousal.
Time Frame: Pre activity
Population: For the Citizen Science group, only 2 (of 3) participants completed the measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 12 | 1 | 1 | 2 | 5 | 2
units on a scale | 14.5 (2.236) | 15 (0) | 16 (0) | 16 (0) | 14 (2.55) | 12.5 (4.95)

13. Primary Outcome: Mood_arousal (Time 2)
Description: Post measures of mood (arousal) was taken using the University of Wales Institute of Science and Technology (UWIST) Mood Adjective Checklist (MACL), an average measure of arousal. The subscale will range from 4 to 16, with higher scores indicating higher arousal.
Time Frame: Post activity (20 minutes after pre-activity measure)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 11 | 1 | 1 | 2 | 5 | 2
units on a scale | 14.64 (1.748) | 16 (0) | 16 (0) | 15 (1.414) | 14.6 (1.673) | 13.5 (3.536)

14. Secondary Outcome: Mobility Limitation
Description: Mobility Limitation was determined using accelerometers to measure participant movement throughout the activities to correlate with physical activity measures.
Time Frame: Throughout activity (measure taken for 20 minutes)
Population: Upon downloading the accelerometer data, we identified technical errors in the recording process. Several accelerometers failed to capture any data, while others recorded data inconsistently, with significant gaps. Due to the incomplete and unreliable nature of the recordings, we determined that the data could NOT be used for analysis. Providing the recorded data will be highly misleading.
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event Data were collected through study completion. Participants may be engaged in up to 3 study visits over 3 weeks. Each visit will be less than 1 hour.
Arm/Group | Citizen Science + Walking + Planting | Citizen Science + Walking | Citizen Science + Planting | Citizen Science | Walking | Planting
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/1 | 0/1 | 0/3 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/1 | 0/1 | 0/3 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 0/12 | 0/1 | 0/1 | 0/3 | 0/5 | 0/2

LIMITATIONS AND CAVEATS:
Study was a pilot, using small samples without comparison groups (such as controls). In addition, the study was a one-off and was unable to explore longer-term studies exploring 'dose' of the activity e.g. longer duration of activity (min), frequency and seasonality effects. Data capture using objective measures (e.g. actual physical exertion rates using accelerometers/mobile health sensors) was unable to be carried out owing to Covid-19 restrictions on direct contact with participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT04913363/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT04913363/ICF_001.pdf